CLINICAL TRIAL: NCT06338995
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Lebrikizumab/LY3650150 in Participants With Chronic Rhinosinusitis With Nasal Polyps on Background Intranasal Corticosteroids
Brief Title: A Study of Lebrikizumab (LY3650150) in Participants With Chronic Rhinosinusitis and Nasal Polyps Treated With Intranasal Corticosteroids (CONTRAST-NP)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18790; J2T-MC-KGBU (Other: Eli Lilly and Company); 2023-508760-29-00 (Other: EU CT Number)
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, parallel group, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lebrikizumab every 2 weeks (Q2W)/ every 4 weeks (Q4W) (Experimental): Lebrikizumab will be given as Subcutaneous (SC) injection. Participants will receive background therapy with intranasal corticosteroids (INCS).
  Note: Enrollment of adolescents will be open-label, with all adolescents assigned to the lebrikizumab Q2W/Q4W treatment arm.
  Interventions: Drug: LY3650150; Drug: Standard therapy for INCS
- Lebrikizumab Q2W/every 8 weeks (Q8W) (Experimental): Lebrikizumab will be given as SC injection. Participants will receive background therapy with INCS.
  Interventions: Drug: LY3650150; Drug: Standard therapy for INCS
- Placebo Q2W/Q4W (Placebo Comparator): Placebo will be given as SC injection. Participants will receive background therapy with INCS.
  Interventions: Drug: Placebo; Drug: Standard therapy for INCS

INTERVENTIONS:
Drug: LY3650150 — Administered SC.
  Arms: Lebrikizumab Q2W/every 8 weeks (Q8W); Lebrikizumab every 2 weeks (Q2W)/ every 4 weeks (Q4W)
Drug: Placebo — Administered SC.
  Arms: Placebo Q2W/Q4W
Drug: Standard therapy for INCS — Administered as intranasal spray.

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of lebrikizumab in participants with chronic rhinosinusitis and nasal polyps treated with intranasal corticosteroids. The study will last about 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed chronic rhinosinusitis (CRS) with bilateral nasal polyps (NP).
* Prior treatment with systemic corticosteroids (SCS) within the last 2 years (or a medical contraindication or intolerance to SCS), prior surgery for NP, or both.
* Endoscopic bilateral NPS score of at least 5 out of 8, with a minimum score of 2 in each nasal cavity performed at screening and baseline.
* Ongoing symptoms for at least 8 weeks prior to study entry (screening), including:

  1. Nasal congestion with moderate or severe symptom severity (score 2 or 3) at screening and a weekly average severity score of at least 1 (range 0 to 3) at randomization, and
  2. At least one other symptom, such as partial loss of smell (hyposmia), total loss of smell (anosmia), or anterior or posterior rhinorrhea.
* Have concomitant asthma must be stable in the 3 months prior to screening using permitted regular asthma treatment.
* Adolescent participants ≥12 to <18 years of age and weighing ≥40 kg at time of Visit 1.

Exclusion Criteria:

* Have received a dose of lebrikizumab.
* Have received treatment with any rescue medication and/or have the need for surgery for NP during screening and/or run-in period.
* Allergen immunotherapy (subcutaneous immunotherapy [SCIT]/sublingual immunotherapy [SLIT]) initiated within 6 months prior to screening, that is not on a stable dose (3 months prior to screening).
* Has received a biologic treatment approved for use in CRSwNP, asthma, or AD, even if administered to treat a different condition, within 4 months or 5 half-lives, whichever is longer, prior to screening.
* Have received treatment with any biologic or systemic immunosuppressants for inflammatory disease or autoimmune disease prior to the baseline visit:

  1. B cell-depleting biologics, including rituximab, within 6 months.
  2. other biologics within 5 half-lives (if known) or 8 weeks, whichever is longer.
  3. Systemic immunosuppressants within 4 weeks prior to baseline.
* Have had any sinus intranasal surgery (including nasal polypectomy) within 6 months prior to screening
* Have had prior sino-nasal surgery or sinus surgery changing lateral wall structure of the nose making it difficult to assess endoscopic NPS
* Have a presence of any of the following conditions that may impact the assessment of endpoints at screening or baseline:

  1. Nasal septal deviation occluding at least one nostril.
  2. Antrochoanal polyps.
  3. Acute sinusitis, acute nasal infection, or acute upper respiratory infection.
  4. Ongoing rhinitis medicamentosa.
  5. Presence of another diagnosis associated with NP (ie, eosinophilic granulomatosis with polyangiitis, granulomatosis with polyangiitis, Young's syndrome, primary ciliary dyskinesia, cystic fibrosis). Note: for adolescents, documentation for ruling out cystic fibrosis and primary ciliary dyskinesia is required.
  6. A nasal cavity tumor (malignant or benign).
  7. Evidence of fungal rhinosinusitis.
* Have anosmia from COVID or any reason other than CRSwNP.
* Participants with forced expiratory volume in 1 second (FEV1) 50% or less (of predicted normal) at screening.
* Female participant who is pregnant, breastfeeding, or is planning to become pregnant, or to breastfeed during the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Mean Change From Baseline (CFBL) in Participant Reported Nasal Congestion Score (NCS) Severity | Baseline, Week 24
  NCS severity is rated by study participants using a 4-point scale (range from 0 to 3), where 0 corresponds to no symptoms and 3 corresponds to severe symptoms. Study participants are asked to record the severity of nasal congestion for the previous 24 hours. This assessment will be collected in the participant eDiary.
Mean CFBL in Endoscopic Nasal Polyp Score (NPS) | Baseline, Week 24
  The endoscopic NPS is assessed by a centralized, blinded, independent review of nasal endoscopy video recordings. The total score is the sum of the right and left nasal cavity scores. For each nasal cavity, endoscopic NPS is graded based on polyp size from 0 to 4, where 0 = no polyps and 4 = large polyps.

SECONDARY OUTCOMES:
Mean change in Opacification of Sinuses Measured by the Lund Mackay score (LMK) | Baseline, Week 24
  Central read on sinus computed tomography (CT) scans for the Lund Mackay score (LMK) will be performed. Review of the CT scans of the right and left frontal sinuses will include the use of a scoring system. The LMK scoring system is a 3-point grading scale where 0 = normal, 1 = partial opacification, and 2 = total opacification. The total score is the sum of the scores from each side and ranges from 0 to 24, where 0 indicates no disease and 24 indicates the most severe disease.
Mean change in Forced Expiratory Volume in 1 Second (FEV1) | Baseline, Week 24
  FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation.
Mean CFBL in Severity of Loss of Smell | Baseline, Week 24
  Participants will be asked about the severity of loss of smell using a 4-point scale, where 0 corresponds to no symptoms and 3 corresponds to severe symptoms. Study participants are asked to record the severity of loss of smell, for the previous 24 hours. This assessment will be collected in the participant eDiary.
Mean CFBL in Postnasal Drip | Baseline, Week 24
  Postnasal drip is rated by study participants using a 4-point scale, where 0 corresponds to no symptoms and 3 corresponds to severe symptoms. Study participants are asked to record the severity of their postnasal drip, at its worst, for the previous 24 hours. This assessment will be collected in the participant eDiary.
Mean Change from Baseline by Visit for the 22-item Sino-nasal Outcome Test (SNOT-22) | Baseline, Week 24
  The 22-item Sino-nasal outcome test assessing sino-nasal and auricular function, psychological impact, productivity, and sleep quality. Participants will be asked to recall their experiences over the past 2 weeks and rate their symptoms on a scale ranging from 0, which corresponds to no problem, to 5, which corresponds to problem as bad as it can be.
Mean Change from Baseline by Visit for the Nasal Peak Inspiratory Flow (NPIF) | Baseline, Week 24
  NPIF measures the maximum inspiratory flow rate through both nostrils during inspiration with results expressed in liters per min (L/min). Participants with NPIF results >120 L/min represent no nasal obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (191):
- United States (34):
  - AllerVie Clinical Research, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Keck Medicine of USC, Arcadia, California
  - University of California, Irvine, Irvine, California
  - DaVinci Research LLC, Roseville, California
  - Breathe Clear Institute, Torrance, California
  - Colorado ENT & Allergy, Colorado Springs, Colorado
  - Orlando ENT & Allergy, Orlando, Florida
  - NuLine Clinical Trial Center, Pompano Beach, Florida
  - University of South Florida, Tampa, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - Entopy Research LLC, Chicago, Illinois
  - Chicago ENT, Chicago, Illinois
  - South Louisiana Ear, Nose, Throat & Facial Plastic Surgery - PPDS, Mandeville, Louisiana
  - Chesapeake Clinical Research, Inc., White Marsh, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Missouri, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Circuit Clinical/Mercer Allergy and Pulmonary Associates, Hamilton, New Jersey
  - Madison ENT & Facial Plastic Surgery, New York, New York
  - New York Allergy and Sinus Center, New York, New York
  - Equity Medical, The Bronx, New York
  - UCMC, Cincinnati, Ohio
  - Optimed Research, LTD, Columbus, Ohio
  - Specialty Physician Associates, Bethlehem, Pennsylvania
  - Medical University of South Carolina- Department of Otolaryngology and Head and Neck Surgery, Charleston, South Carolina
  - Alina Clinical Trials, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas Physicians Department of Otorhinolaryngology Clinc, Houston, Texas
  - Ear Nose and Throat Associates of Texas PA, McKinney, Texas
  - Alamo ENT Associates, San Antonio, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Richmond Ear Nose and Throat, Richmond, Virginia
  - The Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (9):
  - CEMLO - Centro de Especialidades Médicas Lobos, Beunos Aires
  - Fundacion Respirar, Buenos Aires
  - Centro Platense en Investigaciones Respiratorias - CEPIR, Buenos Aires
  - Fundacion CIDEA, Caba
  - Centro de Investigaciones Clínicas - IESR - Rosario, Rosario
  - Investigaciones en Patologías Respiratorias SRL, San Miguel de Tucumán
  - CIMER-Centro Integral de Medicina Respiratoria, San Miguel de Tucumán
  - Centro Respiratorio Infantil, Santa Fe
  - CARE - Centro de Alergia y Enfermedades Respiratorias, Villa Crespo
- Belgium (3):
  - Pneumocare, Erpent
  - UZ Gent, Ghent
  - Cliniques Universitaires Saint-Luc Avenue Hippocrate 10, Woluwe-Saint-Lambert
- Bulgaria (6):
  - Multiprofile Hospital For Active Treatment Dr Tota Venkova A, Gabrovo
  - Medical Center Medconsult Pleven OOD, Pleven
  - Diagnostic-Consultative Centre Ascendent EOOD, Sofia
  - Military Medical Academy - Multiprofile Hospital for Active Treatment - Sofia,, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna, Sofia
  - Multiprofile Hospital for Active treatment Trakia EOOD, Zagora
- Canada (4):
  - St. Joseph's Hospital, Ontario
  - CSAC, Québec
  - The Gordon and Leslie Diamond Health Care Centre, Vancouver
  - St Paul's Sinus Centre, Vancouver
- China (26):
  - Peking University Third Hospital, Beijing
  - Beijing Hospital, Beijing
  - Beijing Tongren Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - The Third Xiangya Hospital of Central South University, Changsha
  - Sichuan Provincial People's Hospital, Chengdu
  - The First People's Hospital of Foshan, Foshan
  - The First Affiliated Hospital Of Fujian Medical University, Fuzhou
  - Shenzhen Second People's Hospital, Guangdong
  - Hainan General Hospital, Haikou
  - Hangzhou First People's Hospital, Hangzhou
  - Huai'an First People's Hospital, Huai'an
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - The first Affilliated Hospital Shandong First Medical University, Shandong
  - Tongji Hospital of Tongji University, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - The First Hospital of Shanxi Medical University, Taiyuan
  - Tianjin People's Hospital, Tianjin
  - Tonghua Central Hospital, Tonghua
  - The 2nd Affiliated Hospital of Wenzhou Medical University, Wenzhou Avenue
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - First People's Hospital of Yinchuan, Yinchuan
- Denmark (4):
  - Aalborg Universitetshospital Medicinerhuset Lungemedicinsk Forskningsenhed, Aalborg
  - Aarhus University Hospital, Dept. of Ear-Nose-Throat, Aarhus
  - Bispebjerg Hospital Department of Respiratory Medicine, Copenhagen
  - Sjællands Universitets Hospital, Køge
- Germany (8):
  - Charite-Universitatsmedizin Berlin, Berlin
  - HNO Zentrum am Kudamm, Berlin
  - Praxis für HNO und Allergologie, Dresden
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - IKF Pneumologie, Frankfurt am Main
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - HNO Praxis, Sachsen
- Hungary (2):
  - Ujpesti Egeszsegugyi Szolgaltato, Budapest
  - Komarom-Esztergom Varmegyei Szent Borbala Korhaz, Tatabánya
- Italy (7):
  - AOU Careggi- University of Florence, Florence
  - Ospedale San Raffaele, Milan
  - AOU Federico II Via Pansini, Napoli
  - Azienda Ospedaliera Di Padova, Padua
  - Azienda Ospedaliero Universitaria Pisana - Stabilimento Santa Chiara, Pisa
  - Fondazione Policlinico A. Gemelli IRCCS, Rome
  - ASST Brianza - Vimercate Hospital, Vimercate
- Japan (35):
  - Toyota Memorial Hospital, Aichi
  - Clinic Kashiwanoha, Chiba
  - University of Yamanashi Hospital, Chūō
  - University of Fukui Hospital, Fukui
  - Saiseikai Fukuoka General Hospital, Fukuoak
  - Matsuda Hospital, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Osaka Habikino Medical Center, Habikino-shi
  - Kansai Medical University Hospital, Hirakata
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital, Hokkaido
  - Hyogo Medical University Hospital, Hyōgo
  - Takarazuka City Hospital, Hyōgo
  - Ibaraki Prefectural Central Hospital, Ibaraki
  - Kagoshima Kouseiren Hospital, Kagoshima
  - Yokohama City Minato Red Cross Hospital, Kanagawa
  - Odawara Municipal Hospital, Kanagawa
  - Tokai University Hospital, Kanagawa
  - Kimitsu Chuo Hospital, Kisarazu
  - 1-8-1, Kishinoura, Kitakyushu
  - 3-54-2, Kotohirahommachi, Kumamoto
  - Kyosai Hospital, Minami-Alps
  - Tohoku Medical and Pharmaceutical University Hospital, Miyagi
  - Ritsuzankai Iida Hospital, Nagano
  - Asahioka, 1-24, Niigata
  - Niigata University Medical & Dental Hospital, Niigata
  - Japan Community Health care Organization Osaka Hospital, Osaka
  - Kansai Electric Power Hospital, Osaka
  - Toho University Sakura Medical Center, Sakura
  - 8-2 Otemachi, Shizuoka
  - Toho University Ohashi Medical Center, Tokyo
  - Nihon University Itabashi Hospital, Tokyo
  - Mie University Hospital, Tsu
  - JCHO Shimonoseki Medical center, Yamaguchi
  - Yamaguchi University Hospital, Yamaguchi
  - Yokohama Minami Kyosai Hospital, Yokohama
- Mexico (5):
  - Avenida Independencia, Aguascalientes
  - Calle Pascual Orozco #2125 col. Magisterial Universidad, Chihuahua City
  - Calle Penitenciaria, Guadalajara Jalsico
  - Miguel Hidalgo 2525, Consultorio 2 Urgencias, Nuevo León
  - Humboldt 302 Col. Centro, Oaxaca City
- Poland (11):
  - Niepubliczny Zakład Opieki Zdrowotnej E-Vita, Bialystok
  - Centrum Medyczne Pratia Katowice, Katowice
  - Centrum Medyczne Angelius Provita, Katowice
  - B&R Clinical Sp. z o.o, Kielce
  - Centrum Medyczne All-Med, Krakow
  - Centrum Medyczne Promed ul. Olszańska 5G, Krakow
  - Specjalistyczny Niepubliczny Zakład Opieki Zdrowotnej Alergologia Plus Ośrodek Diagnostyki, Poznan
  - WIM-PIB, Warsaw
  - Centrum Medyczne Biotamed Morawska Barbara, Wieliczka
  - EMC INSTYTUT MEDYCZNY S.A. Przychodnia, Wroclaw
  - Centrum Medyczne Oporów, Wroclaw
- Portugal (6):
  - Unidade Local de Saúde de Almada-Seixal, E.P.E., Almada
  - ULS da Região de Aveiro, EPE - Hospital Infante D. Pedro, Aveiro
  - Centro Clínico Académico - Braga (2CA-Braga) (Hospital de Braga), Braga
  - Unidade Local de Saúde Loures-Odivelas, Loures
  - ULS do Algarve, EPE - Hospital de Portimão, Seco Portimao Faro
  - Hospital Pedro Hispano, Senhora da Hora
- Romania (5):
  - Centrul Medical Unirea SRL, Brasov
  - Centrul Medical De Diagnostic Si Tratament Ambulator Neomed S.R.L, Brasov
  - Delta Health Care S.R.L, Bucharest
  - Cardiomed S.R.L, Cluj-Napoca
  - Centrul de Excelenta in Rinologie S.R.L, Dolj
- South Korea (10):
  - Inje University Haeundae Paik Hospital, Busan
  - CHA Bundang Medical Center, Gyeonggi-do
  - Pusan National University Hospital, Pusan
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - SNUH - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul
  - Korea University Guro Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Ajou University Hospital, Suwon
- Spain (7):
  - Hospital Universitario Virgen de la Macarena Avenida Dr. Fedriani, Andalucia
  - Centro Médico Teknon, Barcelona
  - Hospital Universitario de Jerez, Cadiz
  - Hospital Clínico Universitario de Santiago, Galícia
  - FutureMeds DKF, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Clinica Universidad de Navarra, Pamplona
- Taiwan (2):
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
- United Kingdom (7):
  - Bristol Royal Infirmary University Hospitals, Bristol
  - Charing Cross Hospital, Chelsea
  - James Paget University Hospitals NHS Foundation Trust, Great Yarmouth
  - Royal Berkshire NHS Foundation Trust, London
  - Guys and St Thomas' NHS Foundation Trust, London
  - Newcastle upon Tyne Hospitals NHSFT Freeman Hospital, Newcastle upon Tyne
  - Stepping Hill Hospital, Stockport

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Lebrikizumab (LY3650150) in Participants With Chronic Rhinosinusitis and Nasal Polyps Treated With Intranasal Corticosteroids (CONTRAST-NP) — https://trials.lilly.com/en-US/trial/472335